CLINICAL TRIAL: NCT04765488
Title: WashIn /WashOut Procedure To Prevent Agitation During Recovery After Inhalational Anesthesia With Sevoflurane: A Multicentral Randomized Trial
Brief Title: WashIn /WashOut Procedure To Prevent Agitation During Recovery After Inhalational Anesthesia With Sevoflurane
Acronym: OPERA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OPERA-001
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Agitation, Emergence; Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: emergence agitation; postoperative agitation; postoperative delirium; postoperative cognitive dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): A group of patients in relation to whom the "Wash In / WashOut" procedure will be applied. In this group we stop the supply of sevoflurane to the first signs of awakening and record the level of sevoflurane , then we resume the supply of sevoflurane to the end-tidal concentration of 1 MAC maintain the anesthesia for 5 min and stop the supply of sevoflurane to the first signs of awakening again, then we resume the supply of sevoflurane to the end-tidal concentration of 1 MAC maintain the anesthesia for 5 min and finally ( the third time) stop supplying sevoflurane and extubate patient after recovery of muscle tone, spontaneous breathing and consciousness.
  Interventions: Procedure: WashIn /WashOut
- Control group (No Intervention): A group of patients in relation to whom will be applied the traditional method of recovery from anesthesia. In this group during the period of awakening we stop supplying sevoflurane and extubate patient after recovery of muscle tone, spontaneous breathing and consciousness.

INTERVENTIONS:
Procedure: WashIn /WashOut — According "Wash In / WashOut" procedure in study group we stop the supply of sevoflurane to the first signs of awakening and record the level of sevoflurane , then we resume the supply of sevoflurane to the end-tidal concentration of 1 MAC maintain the anesthesia for 5 min and stop the supply of sevoflurane to the first signs of awakening again, then we resume the supply of sevoflurane to the end-tidal concentration of 1 MAC maintain the anesthesia for 5 min and finally ( the third time) stop supplying sevoflurane and extubate patient after recovery of muscle tone, spontaneous breathing and consciousness.
  Arms: Study group

SUMMARY:
Inhalation anesthesia is the most frequently used technique and is performed in around 70% of surgeries worldwide. Sevoflurane is the most frequently used halogenated anesthetic and is used in 2/3 of the cases.

The anesthetic strength of inhalation agents was established in the classic work of Eger and colleagues who determined the minimum alveolar concentration (MAC) of an inhaled anesthetic at atmospheric pressure, necessary to prevent a motor reaction in response to a pain stimulus in 50% of patients.

Agitation is a frequent anesthesia complications and it not only lengthens the period of post anesthetic awakening and need for advance monitoring of the patient, but may be a predisposing factor in the development of postoperative delirium (POD) and postoperative cognitive dysfunction (POCD) which are independent predictors of increased mortality, prolonged treatment in the ICU and hospital, and prolonged social adaptation of the operated patients.(The ability of the patient to serve themselves independently.).

There is a fairly popular point of view that there is no specific prophylaxis or treatment of postoperative agitation.

However, a variant of anesthesia induction with sevoflurane was recently proposed, which reduced the frequency of agitation in children from 24.7% to 4.4%. The technique consisted in interrupting anesthesia at the moment of loss of consciousness, awakening the patient and subsequently performing re-induction. Since this technique might be time consuming in the busiest period of a surgical theatre and not safe if performed with the airways still unsecured it is advisable to shift the Wash In/Wash Out procedure to the stage of awakening at the end of surgery.

DETAILED DESCRIPTION:
Inhalation anesthesia is the most frequently used technique and is performed in around 70% of surgeries worldwide. Sevoflurane is the most frequently used halogenated anesthetic and is used in 2/3 of the cases.

The anesthetic strength of inhalation agents was established in the classic work of Eger and colleagues who determined the minimum alveolar concentration (MAC) of an inhaled anesthetic at atmospheric pressure, necessary to prevent a motor reaction in response to a pain stimulus in 50% of patients. Since alveolar concentrations of inhaled anesthetics correspond to their concentrations in other organs after equilibrium, which is most quickly achieved in organs with rich perfusion, such as the brain and heart, MAC is an analogue of the plasma EC50 (concentration effective at 50%) for intravenous anesthetics. 1 MAC of sevoflurane is equal to an end-tidal concentration of 2.0 volume percent.

Agitation is a frequent anesthesia complications and it not only lengthens the period of post anesthetic awakening and need for advance monitoring of the patient, but may be a predisposing factor in the development of postoperative delirium (POD) and postoperative cognitive dysfunction (POCD) which are independent predictors of increased mortality, prolonged treatment in the ICU and hospital, and prolonged social adaptation of the operated patients.(The ability of the patient to serve themselves independently.).

Despite the fact that attempts to reduce the risk of postoperative neurological complications have been made repeatedly, the frequency of occurrence of agitation in the early post operative period in adult patients is up to 30%.

Some authors drew attention to the need to comply with the basic requirements for the safety of anesthesia: continuity and adequacy of anesthesia, and avoidance of excessively deep or too superficial level of anesthesia. Other authors consider it suitable to use midazolam, propofol, opioid and non-opioid analgesics in case of agitation. Magnesium and calcium chloride were also tested to stop the described phenomenon, but their beneficial effects were not confirmed in subsequent investigations.

There is a fairly popular point of view that there is no specific prophylaxis or treatment of postoperative agitation.

However, a variant of anesthesia induction with sevoflurane was recently proposed, which reduced the frequency of agitation in children from 24.7% to 4.4%. The technique consisted in interrupting anesthesia at the moment of loss of consciousness, awakening the patient and subsequently performing re-induction. Since this technique might be time consuming in the busiest period of a surgical theatre and not safe if performed with the airways still unsecured it is advisable to shift the Wash In/Wash Out procedure to the stage of awakening at the end of surgery. The authors also have occasionally experienced high quality awakenings in patients who received this technique, without side effects or patients' discomfort.

Objective: The primary objective for the multicentral OPERA Trial will be to explore the effect of the "Wash In / WashOut" procedure at the end of the operation on the incidence of post-anesthetic agitation, delirium and postoperative cognitive dysfunction.

Treatment groups

All patients undergoing non-cardiac surgery under general inhalation anesthesia will be randomly assigned to one of two groups.

1. Control group.

   A group of patients in relation to whom will be applied the traditional method of recovery from anesthesia. In this group during the period of awakening, the supply of sevoflurane will be stopped and the patient will be extubated after recovery of muscle tone, spontaneous breathing and consciousness.
2. Investigating group.

   A group of patients in relation to whom the "Wash In / WashOut" procedure will be applied. In this group the supply of sevoflurane will be stopped to the first signs of awakening and record the level of sevoflurane , then the supply of sevoflurane will be resumed to the end-tidal concentration of 1 MAC maintain the anesthesia for 5 min and stop the supply of sevoflurane to the first signs of awakening again, then the supply of sevoflurane will be resumed to the end-tidal concentration of 1 MAC maintain the anesthesia for 5 min and finally ( the third time) stop supplying sevoflurane and extubate patient after recovery of muscle tone, spontaneous breathing and consciousness.
3. Perioperative and anesthetic management

Intraoperative monitoring will include continuous assessment of hemodynamic parameters (NIBP, ECG), SpO2, analysis of expiratory gases (CO2, O2, sevoflurane), ABB analysis of arterial or mixed venous blood(for patients (from both group)whose monitoring indicators during surgery ( saturation ) will go beyond the reference values ( less than 95 % )). Benzodiazepines, ketamine, , antipsychotics should not be used in premedication, induction, and while maintaining anesthesia.

In both groups, induction is achieved by intravenous administration of propofol, to patients under the age of 55 at a dosage of 2 mg / kg of ideal body weight until they lose consciousness, to patients older than 55 years and to patients of classes III and IV according to ASA 1 mg / kg ideal body weight until unconscious, with fentanyl at a dose of 2-3 μg / kg or mask induction with sevoflurane 2 l / min 3 MAC with fentanyl at a dosage of 4 μg / kg.

Maintenance of anesthesia in both groups is ensured by the use of sevoflurane with a finite alveolar concentration 1 MAC and fentanyl (0.05-0.1 mg as needed, according to the decision of the attending anesthesiologist). Muscle relaxants(monitoring of curarization and reversal will not be carried out) , vasoactive drugs, infusion solutions, adjuvants, with the exception of those listed above (if there is no strict need for them), are selected at the discretion of the anesthesiologist.

During the awakening period, the time from the sevoflurane interruption until the occurrence of spontaneous breathing, the time before opening the eyes, the time before extubation, the time before orientation is recorded. The criterion of awakening the patient will be considered the ability to perform the simplest commands: open your eyes, raise your head, show your tongue. The patient is assessed on the RASS scale immediately after awakening, 15 minutes after awakening and 30 minutes after awakening.

After awakening, assessing severity of the condition, the need for prolonged mechanical ventilation, vasopressor or inotropic support, the need for monitoring in ICU, the patient is transferred to the unit or to ICU (The Aldrete Scale will be used to assessment of the patients condition) , where he will be monitored for hemodynamics (NIBP, ECG, SpO2), a dynamic assessment of the general state, monitoring of laboratory parameters and postoperative therapy, according to current practice.

Preoperative examination, anesthesia management, pre- and postoperative therapy will be carried out in accordance with current practice. All data from laboratory and instrumental assessments, as well as all medical documentation (protocol of anesthesia course, anesthesia card, patient management cards in the ICU, prescriptions) will be available as part of the clinical study to treating doctor.

Trial Mechanics, Methodology, & Analysis

The following measures will allow us to achieve a high level of protocol adherence in this trial: research teams will be created in each participating hospital, which will consist of anesthesiologists and nurse anesthetists. Each research team will be responsible for conducting a "Wash In / WashOut" procedure to each randomized patient. All members of the research team will be instructed on the technique of "WashUp / WashOut" procedure before the start of the study. All the data obtained in this study will be recorded in medical documentation (protocol of anesthesia course, anesthesia card, patient management cards in the ICU, prescriptions) and patient's case report forms.

Statistical analysis

The frequency of the primary endpoint was considered and the relative reduction was associated with sequential awakening by sevoflurane. Considering a type I error of 0.05 and a power of 80% (type II error of 0.2), the required number was 98 patients per group. Planned to enroll 100 patients in each groupsurgery study arm to account for possible dropouts. 200 patients summary.

All data will be analyzed according to the intention-to-treat principle. No imputation will be applied for missing data. Per-protocol analyses will be also performed. Demographic and baseline disease characteristics will be summarized with the use of descriptive statistics. Categorical variables will be reported as absolute numbers and percentages. Unadjusted univariate analyses, to compare the two treatment groups, will be based on Chi-square or Fisher's exact test. Relative risks and 95% confidence intervals will be calculated by means of the two-by-two table method with the use of log-normal approximation. Continuous variables will be reported as mean ± standard deviation (SD) or median and interquartile range (IQR). Between-group differences will be evaluated using the t-test or Wilcoxon signed rank test, in accordance with normality of the distribution.

A logistic regression model using a stepwise selection will be used to estimate the treatment effect and predictors of primary endpoint. The pre-randomization clinical data and center will be entered into the model if their univariate p value is< 0.1 and there is no correlation between them. Collinearity and overfitting will be assessed using a stepwise regression model and Pearson correlation test. The treatment group will be forced into the multivariate model.

An independent safety committee will perform three interim analyses after recruitment of 25%, 50% and 75% of patients. Data evaluation at each interim analysis will be based on the alpha spending function concept, according to Lan and De Mets', and will employ O'Brien-Fleming Z-test boundaries, which are very conservative early in the trial. For the first interim analysis the efficacy stopping rule would require an extremely low p value (p < 0.000015). For the second interim analysis p < 0.003 will be taken as efficacy stopping rule. For the third interim analysis p < 0.02 will be taken as efficacy stopping rule. Investigators will be kept blind to the interim analysis results.

The Data Safety and Monitoring Committees will also perform conditional power analyses in order to evaluate potential interruption for futility issues in the trial. Conditional power will be calculated by assuming that the proportion of outcomes will follow the observed trend.

The following analysis will be performed to determine the effect of sequential awakening by sevoflurane on different subgroups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from participants
2. Age ≥ 18 years
3. Planned open abdominal surgery
4. General anesthesia

Exclusion Criteria:

1. Pregnant patients and breastfeeding patients
2. Mental disorders
3. Epilepsy, Parkinson disease, Alzheimer, peripheral nerve and neuromuscular junction pathology (amyotrophic lateral sclerosis, Guillain-Barre Syndrome, myasthenia gravis et cet.)
4. Use of antidepressants, antipsychotics, sedatives, psychoactive drugs within a month before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
The effect of "Wash In / WashOut" procedure on the incidence of postoperative agitation after anesthesia with sevoflurane. | during 30 minutes after awaking
  the patient scores +2 or more points on the RASS scale in one or more measurements, then he is diagnosed with agitation.
To estimate changes in the incidence of postoperative agitation on the RASS scale | during 30 minutes after awaking
  incidence of postoperative agitation in control group - incidence of postoperative agitation in study group

SECONDARY OUTCOMES:
To estimate changes in the incidence of postoperative delirium on the scales CAM-ICU, ICDSC | 3 days after surgery twice a day (a.m. and p.m.)
  incidence of postoperative delirium in control group - incidence of postoperative delirium in study group
To estimate changes in the incidence of postoperative cognitive impairment | on the 7th day after surgery
  incidence of postoperative cognitive impairment in control group - incidence of postoperative cognitive impairment in study group
To estimate the incidence of postoperative nausea and vomiting, the need of using of antiemetics | Since end of surgery prior to hospital discharge
  incidence of postoperative nausea and vomiting, the need of using of antiemetics in control group - incidence of postoperative nausea and vomiting, the need of using of antiemetics in study group
To estimate patient satisfaction with anesthesia on the ISAS scale | At third postoperative day
  Result of The Iowa Satisfaction with Anesthesia Scale (ISAS)
Length of stay in ICU | ICU discharged
  The date of ICU discharged - the date of surgery
The duration of hospitalization | Hospital discharged
  The date of hospital discharged - the date of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University); Head of Research V. Negovsky Reanimatology Research Institute; Giovanni Landoni, Study Chair — San Raffaele Scientific Institute; Pavel Bagdasarov, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (3):
- Russia (3):
  - Moscow Scientific Clinical Center, Moscow
  - Moscow Regional Research and Clinical Institute Moniki n.a. M.F. Vladimirskiy, Moscow
  - Clinical hospital №1 of the I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow

IPD SHARING:
Plan to Share IPD: No
Our Local Ethical Committee disable us to do it